CLINICAL TRIAL: NCT05260320
Title: Anesthetic Optimization in Pediatric LeFort Surgeries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00316335
Record Dates: First submitted 2022-02-02; First posted 2022-03-02 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Le Fort; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: All consented patients will receive the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Standardized Protocol (Experimental): Preop considerations
  1. Ensure CBC, PT, PTT, type and cross are available, if not obtain with preop IV access
  Premed
  1. Acetaminophen PO 15mg/kg
  2. Scopolamine patch as indicated
  3. Midazolam as indicated PO or IV
  Induction
  1. Standard induction with lidocaine (1.5 mg/kg), propofol (1-3 mg/kg), and rocuronium (0.6mg/kg)
  2. Fentanyl 100 mcg bolus
  3. Dexmedetomidine 0.3 mcg/kg bolus
  4. Nasotracheal intubation (NTI) - surgical team will suture to nasal septum
  5. Place an additional PIV, ideally large gauge for volume resuscitation (18g or 16g)
  6. Dexamethasone 4-8mg q4-6 hours per surgical request
  7. Tranexamic acid 30mg/kg bolus (over 15 minutes)
  8. Ancef 30 mg/kg bolus
  Monitors /Access
  1. Standard ASA monitors
  2. Avoid placing nasal or oral temperature probe as this interferes with surgical exposure
  3. PIV x 2 is sufficient, have at least one large gauge PIV for volume resuscitation
  4. Arterial catheter not necessary but place as needed, especially if patient is medically compl
  Interventions: Other: Standardized Anesthetic Course from Premedication to Induction

INTERVENTIONS:
Other: Standardized Anesthetic Course from Premedication to Induction — See information in intervention group description

SUMMARY:
This study will propose and evaluate a standardized LeFort osteotomy anesthetic protocol for pediatric patients at Johns Hopkins Hospital. There are two cohorts to this study: a prospective cohort who will receive the study anesthesia protocol and a historical cohort that received standard of care. The investigators hope this will help to minimize unnecessary postoperative pain management, inpatient stay, and long-term morbidity and mortality in these patients.

DETAILED DESCRIPTION:
This study will propose and evaluate a standardized LeFort osteotomy anesthetic protocol for pediatric patients at Johns Hopkins Hospital. There are two cohorts to this study: a prospective cohort who will receive the study anesthesia protocol and a historical cohort that received standard of care. The investigators hypothesize that implementation of this standardized protocol will show improved surgical outcomes among these patients as compared to current (discretionary) treatment. This study aims to optimize the anesthetic management of these patients in order to minimize postoperative pain management, inpatient stay, and long-term morbidity and mortality in these complex patients.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing Le Fort osteotomy at Johns Hopkins Hospital
* Age >= 14 years

Exclusion Criteria:

* Contraindications to standardized anesthetic protocol (intervention arm)

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | From hospital admission (on day of surgery) to discharge, which is expected to last 2-7 days though may be up to 30 days
  The degree (as ranked on a scale from 1-10) and duration of postoperative pain, including necessity of postoperative analgesia

SECONDARY OUTCOMES:
Length of stay | From hospital admission (on day of surgery) to discharge, which is expected to last 2-7 days though may be up to 30 days
  Length of inpatient stay (in days)
Critical care utilization | From hospital admission (on day of surgery) to discharge, which is expected to last 2-7 days though may be up to 30 days
  Utilization, and, where appropriate, length of use of the following: ICU, ventilatory support, intubation, blood products

CONTACTS AND LOCATIONS:
Overall Officials: Robin Yang, MD, DDS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with those conducting research data collection and analysis, and IPD that underlie results in a publication will be published.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will become available to the study team upon collection and will be deleted after publication
Access Criteria: IPD access will be granted to those researchers making significant contributions to data collection or analysis, at the discretion of the principal investigator

REFERENCES:
- [Background] SADOVE MS. Anesthetic management for maxillofacial surgery. Ill Med J. 1956 Nov;110(5):227-31. No abstract available. PMID 13376109
- [Background] Lucin Yagual TA, Vivanco Murillo SM, Espinoza Daquilema NV, Mariscal Garcia RS, Dick Paredes DF. Smooth Extubation Techniques in Pediatric Patients After LeFort I Osteotomy. Cureus. 2021 Apr 24;13(4):e14659. doi: 10.7759/cureus.14659. PMID 34046286
- [Background] Krishna SG, Bryant JF, Tobias JD. Management of the Difficult Airway in the Pediatric Patient. J Pediatr Intensive Care. 2018 Sep;7(3):115-125. doi: 10.1055/s-0038-1624576. Epub 2018 Jan 28. PMID 31073483
- [Background] Gleizal A, Di Rocco F, Chauvel-Picard J. Indications of Lefort osteotomies for facial deformities induced by craniosynostosis. Neurochirurgie. 2019 Nov;65(5):279-285. doi: 10.1016/j.neuchi.2019.10.002. Epub 2019 Oct 16. No abstract available. PMID 31645264
- [Background] Tewari A, Singh G, Mishra M, Gaur A, Mallan D. Comparative Evaluation of Hypotensive and Normotensive Anesthesia on LeFort I Osteotomies: A Randomized, Double-Blind, Prospective Clinical Study. J Maxillofac Oral Surg. 2020 Jun;19(2):240-245. doi: 10.1007/s12663-019-01325-7. Epub 2020 Jan 17. PMID 32346234
- [Background] Wong GB, Nargozian C, Padwa BL. Anesthetic concerns of external maxillary distraction osteogenesis. J Craniofac Surg. 2004 Jan;15(1):78-81. doi: 10.1097/00001665-200401000-00022. PMID 14704568
- [Background] Posnick JC, Choi E, Chavda A. Operative Time, Airway Management, Need for Blood Transfusions, and In-Hospital Stay for Bimaxillary, Intranasal, and Osseous Genioplasty Surgery: Current Clinical Practices. J Oral Maxillofac Surg. 2016 Mar;74(3):590-600. doi: 10.1016/j.joms.2015.07.026. Epub 2015 Aug 5. PMID 26303951
- [Background] Lopez MM, Zech D, Linton JL, Blackwell SJ. Dexmedetomidine Decreases Postoperative Pain and Narcotic Use in Children Undergoing Alveolar Bone Graft Surgery. Cleft Palate Craniofac J. 2018 May;55(5):688-691. doi: 10.1177/1055665618754949. Epub 2018 Feb 15. PMID 29446987
- [Background] Precious DS, McFadden LR, Fitch SJ. Orthognathic surgery for children. Analysis of 88 consecutive cases. Int J Oral Surg. 1985 Dec;14(6):466-71. doi: 10.1016/s0300-9785(85)80051-x. PMID 3936793